CLINICAL TRIAL: NCT00761917
Title: Analysis of the Tear Film Lipid Layer
Brief Title: Diagnostic Evaluation of the Tear Film
Status: Completed | Type: Observational
Sponsor: TearScience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: KS010
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Normal: Subjects without dry eye symptoms based on questionnaire.
  Interventions: Device: Tear Film Analyzer
- 2: Dry Eye: Subjects with dry eye symptoms based on questionnaire.
  Interventions: Device: Tear Film Analyzer

INTERVENTIONS:
Device: Tear Film Analyzer — tear film images
  Other Names: ocular surface interferometry

SUMMARY:
The objectives of this study are to assess for a difference between normal and dry eye subjects in tear film quality using a diagnostic interferometry device and to determine whether there are associations between tear film quality and dry eye symptoms and signs.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 year of age or older
* Willing and able to comply with study exam procedure

Exclusion Criteria:

* Eyelid abnormality or ocular surface condition affecting ability to visualize tear film
* Women who are pregnant or nursing
* Any of the following conditions within specified timeframe prior to study participation:

  1. Instillation of eye drops
  2. Contact lens wear
  3. Use of oil-based facial cosmetics
  4. Swimming in chlorinated pool
  5. Eye examination procedures that may affect the tear film
  6. Participation in another ophthalmic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing routine eye examination in ophthalmic practices
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Tear film analysis of lipid layer quality | upon enrollment

SECONDARY OUTCOMES:
Dry Eye Symptoms | upon enrollment
Tear Film Break-Up Time | upon enrollment
Corneal and Conjunctival Staining | upon enrollment
Meibomian Gland Assessment | upon enrollment
Schirmer Test | upon enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Christy Stevens, OD, Study Director — Kolis Scientific
Locations (8):
- United States (8):
  - Fayetteville, Arkansas
  - Morrow, Georgia
  - Oak Lawn, Illinois
  - Edgewood, Kentucky
  - Bloomington, Minnesota
  - Chesterfield, Missouri
  - Charlotte, North Carolina
  - Henderson, North Carolina